CLINICAL TRIAL: NCT00127374
Title: Mood and Behavior Changes Among Overweight Adolescent Females
Status: Withdrawn | Type: Observational
Why Stopped: withdrawn due to non-response. PI left university
Sponsor: University of Kentucky (Other)
Other Study IDs: 04-0541-F3R
Record Dates: First submitted 2005-08-04; First posted 2005-08-05 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Obesity; Depression
Keywords: Overweight; self-esteem; depression
MeSH Terms: conditions — Obesity; Depression; Overweight | interventions — Diet

INTERVENTIONS:
Behavioral: Dietary and physical activity modifications

SUMMARY:
The specific aims of this study are to document the co-existence of depression, low self-esteem, and high-risk behaviors among overweight and at-risk for overweight female adolescents; and decrease the prevalence of high-risk behaviors by improving depressive symptoms/signs and self-esteem through weight management intervention strategies that encourage long-term mental and physical well being. The proposed research will test the following hypotheses:

* Overweight and at-risk for overweight female adolescents have poor self-esteem that may mask depression and mediate high-risk behaviors; and
* Improved weight perception decreases participation in high-risk behavior secondary to improved self-esteem and depression.

DETAILED DESCRIPTION:
How adolescents view (self-concept) and value themselves (self-esteem) may predict future adjustment and success in life. Self-concept comprises assessment of scholastic, athletic and job competence, social acceptance, physical appearance, romantic appeal, behavioral conduct, close friendship, and global self-worth. Self-esteem is the feeling of self-acceptance, goodness, and worthiness. It influences daily activities, motivation and behavior.

Adolescents are very vulnerable to low self-esteem. Generally, boys have higher self-esteem than girls; higher weight students have lower self-concept; and post-menarcheal females have the poorest opinion of their physical appearance. Higher body mass index (BMI) predicts more negative self-concept. Body image and physical appearance contribute to general physical self-concept and self-esteem.

Regardless of race, gender, age, and socioeconomic status individuals are discriminated against on the basis of weight. Weight-based stigmatization influences self-perception and the perceptions of significant others. Sustained low self-esteem may precipitate anxiety, depression, under achievement, poor motivation and inadequate interpersonal relations.

Obese adolescents are stigmatized by peers. They may attempt to protect their self-image by participating in high-risk behaviors. Obese adolescent girls are more likely to report adverse social, educational and psychological correlates than obese boys. Overweight girls, but not overweight boys, manifest more depressive symptoms than their normal-weight peers. Gender differences in clinical depressive syndromes may emerge in early childhood as opposed to puberty as previously thought.

Early stigmatization of obese children may explain their lower self-esteem and greater shame, humiliation, and perceived teasing compared with their nonobese peers. Studies have found increased psychopathology among clinical samples of obese children and demonstrated improvements in psychological functioning with weight loss. Implementing lifestyle changes during early adolescence, ages 10 to 13 years, and middle adolescence, ages 14 to 16 years, may hold the key for preventing obesity and depression.

The study population will consist of approximately 100 overweight or at-risk for overweight female volunteers, 10 - 14 years old.

ELIGIBILITY:
Inclusion Criteria:

* Girls 10 through 14 years of age who are in good general health and have a BMI in the 85th to 95th percentile or greater than the 95th percentile
* Availability of a parent or guardian to ensure the child attends all monthly clinic visits and who will be available to attend the monthly educational sessions if the child is assigned to the intervention group

Exclusion Criteria:

* Cardiac or pulmonary conditions such as cystic fibrosis, congenital heart disease, or other conditions that would impair ability to do fitness testing
* Physical challenges such as deformities that would impair ability to perform physical activities
* Use of medications such as corticosteroids, seizure medication, or other central nervous system (CNS) medications that would interfere with daily physical activity

Ages: 10 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2005-01; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Decreased body mass index; increased physical activity

SECONDARY OUTCOMES:
Improved self-esteem; improved depression scale score; decreased risk-taking behavior

CONTACTS AND LOCATIONS:
Overall Officials: Joan R Griffith, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States